CLINICAL TRIAL: NCT00979511
Title: The Effect of a 10-month School-based Provision of High-calcium Milk and Weight-bearing Exercise Program on the Bone Mineral Status of 7 to 9 Year Old Pre-pubertal Girls
Brief Title: Effect of High-Calcium Milk and Weight-Bearing Exercise on Bone Mineral Status of Pre-Pubertal Girls
Acronym: Bone Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutrition Center of the Philippines (Other)
Collaborators: Nestlé Foundation (Other)
Responsible Party: Principal Investigator, Cherry C. Maramag, Research Scientist, Nutrition Center of the Philippines
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2009-01
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Osteoporosis
Keywords: osteoporosis; calcium; weight-bearing exercise; bone mass; prepubertal girls
MeSH Terms: conditions — Osteoporosis | interventions — Milk; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 Hi-Calcium milk & exercise (Experimental)
  Interventions: Other: milk and exercise
- 2 Hi-calcium milk with passive exercise (Experimental)
  Interventions: Other: milk and exercise
- 3Low-Calcium with exercise (Experimental)
  Interventions: Other: milk and exercise
- 4 Low-calcium milk with passive exercise (Experimental)
  Interventions: Other: milk and exercise

INTERVENTIONS:
Other: milk and exercise — * milk fortified with 1000mg calcium or low-calcium milk
  * weight-bearing exercise or passive exercise

SUMMARY:
Osteoporosis has been described as a paediatric disease with a geriatric outcome. This is because bone mass is acquired during youth and is progressively lost later in life, without symptom or pain, until a fracture occurs. The proper management of osteoporosis includes improving bone mineral content in the first two decades of life so that reserves are built up before bone loss ensues.

The investigators aim to determine the effect of a 10-month school-based provision of high-calcium milk and weight-bearing exercise program on the bone mineral status among prepubertal girls. The investigators' study is novel since it seeks to determine the effect of these interventions in girls, whose overall risks are much higher for osteoporosis later in life, and in a developing country population whose calcium intakes are more likely to be depleted.

The investigators hypothesize that provision of either high-calcium milk or weight-bearing exercises will improve bone mineral density among prepubertal girls but that the bone accrual will be greater among those with both interventions. In addition, the investigators hypothesize that the changes will be more marked among those whose calcium intakes are lower.

This study will use a two-by-two factorial design of 1) high-calcium milk (1000 mg/day) vs. placebo (115 mg/day) and 2) weight-bearing exercises (a total of 90 to 150 minutes per week divided into 3 to 5 schooldays) vs. no-exercise (passive activities) in a randomized controlled trial, for a total of 4 intervention groups: calcium+exercise, placebo+exercise, calcium+no exercise, placebo+no exercise.

The study will be conducted among 80 prepubertal girls (on Tanner stage 1), aged 7-9 years and enrolled in one primary school in one of the metropolitan cities in the Philippines with an institution or a hospital with a Lunar Prodigy Central dual-energy x-ray absorptiometry (DEXA) machine.

Osteoporosis has no treatment. The problem will continue to become burdensome in the future since population aging per se will increase the risk and incidence of fractures. Understanding the relationship between calcium and exercise is important since the greatest benefit is in the paediatric age range. The study results could provide information on a workable intervention that promotes the multiple health benefits of both exercise and high-calcium milk to young children.

ELIGIBILITY:
Inclusion Criteria:

* pre-pubertal girls on Tanner stage 1
* enrolled in study school
* no diagnosed disorders
* not taking medications that affects bone metabolism or weight-bearing exercise

Exclusion Criteria:

* not meeting the inclusion criteria

Ages: 7 Years to 9 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
bone mass | at baseline, at 5 months, at post-intervention

SECONDARY OUTCOMES:
bone area | at baseline, at 5 months, at post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pura R Solon, MD, Principal Investigator — Clinical Research Scientist
Locations (1):
- Public school, Manila, Manila, Philippines